CLINICAL TRIAL: NCT03675386
Title: Ontario Transitional Pain and Opioid Safety Program: Improving Pain and Opioid Practices for Complex Chronic Pain Patients Following Surgery
Brief Title: Reducing Opioid Use for Chronic Pain Patients Following Surgery
Acronym: RECOUP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-5207
Record Dates: First submitted 2018-05-11; First posted 2018-09-18 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Chronic Pain; Opioid Use; Postoperative Pain; Opioid Dependence
MeSH Terms: conditions — Chronic Pain; Pain, Postoperative; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients in the control group will receive standard care, which involves standard postoperative follow-up with their surgeon/primary care provider. Patients will also be sent with a link for an online multimedia tool during each follow-up time point that will provide information and education regarding non-pharmacologic techniques for managing pain. At the end, all patients in the control arm will be invited to join the TPSP after one year of follow-up if they are still taking opioids.
  Interventions: Other: Control Intervention
- Interventional Group (Experimental): Patients in the interventional group will be given a Transitional Pain Service follow-up appointment at the following postoperative time points (2 to 6 visits for the first two months, and then 1 to 2 visits on a monthly basis until one year). At each visit, patients will meet with the clinical psychologist and chronic pain specialist. Patients in the intervention group will have access to the Manage My Pain (MMP) App. which allows people living with pain to quickly and easily track their pain and function on a daily basis on their smartphones or a browser on their desktop or mobile device. One-page clinical reports will capture the changes in patients' outcome data between clinical visits over the course in time.Clinic visits can be offered in person at the hospital or over telehealth (video conference) based on the patient's preference and clinician's judgment for telehealth suitability.
  Interventions: Other: Interventional Group

INTERVENTIONS:
Other: Interventional Group — The Transitional Pain Service Program enables targeted, mechanism-based, treatment innovations aimed at reducing the incidence and severity of chronic post-surgical pain, disability and enabling safe opioid prescribing/ weaning after major surgery. The investigator's TPSP intervention uses a variety of methods to support patients to manage pain and wean off opioids. This includes physician-guided opioid and non-opioid pharmacotherapy and tapering, and clinical psychology services specializing in pain education, Acceptance & Commitment Therapy (ACT) and e-mobile self-management tools.
  Other Names: Transitional Pain Service Program
  Arms: Interventional Group
Other: Control Intervention — Patients in the control group will receive standard care, which involves standard postoperative follow-up with their surgeon/primary care provider. Patients will also be sent with a link for an online multimedia tool during each follow-up time point that will provide information and education regarding non-pharmacologic techniques for managing pain. At the end, all patients in the control arm will be invited to join the TPSP after one year of follow-up if they are still taking opioids.
  Arms: Control Group

SUMMARY:
Patients with chronic pain are often prescribed long-term opioid therapy, despite the serious risks and growing concerns related to opioid use. The Toronto General Hospital has created the world's first multidisciplinary perioperative Transitional Pain Service Program (TPSP) aimed at reducing the incidence and severity of chronic post-surgical pain. The TPSP incorporates a variety of mechanisms and interventions to help patients manage pain and to wean off opioids. The approach consists of: pain education, Acceptance and Commitment Therapy (ACT), and an e-mobile self- management tool to help patients manage chronic pain more effectively. With the TPSP team, the investigators hope to continually assist patients to achieve a balance between the benefits and potential harms of opioid use to promote long-term health and well-being.

DETAILED DESCRIPTION:
The proposed research program encompasses several study designs to evaluate the effectiveness and potential implementation of the TPSP across Ontario. The investigators will use three approaches to create a comprehensive evidence-base that can be used to guide future policy and programs related to the management of surgical patients with complex pain and chronic opioid use. In the first phase, a multicenter randomized controlled trial will be conducted in 6 hospital sites to evaluate the effectiveness and potential implementation of TPSP across Ontario. The aim is to recruit a total of 210 patients who are currently taking opioids and also undergoing a surgical intervention. The randomized controlled trial will determine the effectiveness of the TPSP at weaning patients completely off opioids while still managing pain after one year. Secondly, an economic and healthcare utilization analysis of the program via linkage to provincial administrative databases will be carried out to understand the impact the TPSP program has on the healthcare system as a whole. Lastly, a qualitative study will be conducted on both the treatment and control groups. The investigators hope to capture further insight to understand patients and providers experiences of the TPSP intervention.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Taking 20 -- 200 mg of preoperative oral morphine equivalents daily
* Any type of surgical procedure, with the exception of those with palliative intent or organ transplantation
* Able to read and understand English as posed on the questionnaire surveys prior to informed consent
* Must be taking opioids for at least one month prior to their operation
* Must have a personal email address for the set-up of the Manage My Pain (MMP) App or online multimedia tool

Exclusion Criteria:

• Subjects who are undergoing palliative care or procedures, organ transplantation, or prescribed with Methadone/Buprenorphine will be excluded from the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2018-09-24 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Portion of patients weaned off opioids | 1 year
  Opioid weaning measured by number of patients successfully weaned off opioids comparing the intervention arm versus control arm
Pain interference | One year
  Brief Pain Inventory Scale is a measure that assess the severity of pain and the impact of pain on daily functions. Measurement of this scale is rated on a 0-10 numerical-rating-scale ( 0= No Pain to 10= Pain as bad as you can imagine or 0= Does not interfere to 10= Completely interferes). The BPI assess pain at its worst, least, average, and now. Pain Severity Score is calculated by adding the scores for questions 2, 3, 4 and 5 and then dividing by 4. This gives a severity score out of 10. Pain Interference Score is calculated by adding the scores for questions 8a, b, c, d, e, f and g and then dividing by 7. This gives an interference score out of 10.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Ladha, MD, Principal Investigator — Toronto General Hospital, University Health Network; Hance Clarke, MD, PhD, Principal Investigator — Toronto General Hospital, University Health Network; Elaheh Adly, MD, Principal Investigator — Hamilton Health Sciences Centre; Paul Tumber, MD, Principal Investigator — University Health Network, Toronto; Anton Marinov, MD, Principal Investigator — Rouge Valley Medical Centre; Melanie Toman, MD, Principal Investigator — Thunder Bay Reginal Health Sciences Centre; Yuvaraj Kotteeswaran, MD, Principal Investigator — Thunder Bay Reginal Health Sciences Centre; Duminda Wijeysundera, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- Toronto General Hospital- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angst MS, Clark JD. Opioid-induced hyperalgesia: a qualitative systematic review. Anesthesiology. 2006 Mar;104(3):570-87. doi: 10.1097/00000542-200603000-00025. PMID 16508405
- [Background] Fletcher D, Martinez V. Opioid-induced hyperalgesia in patients after surgery: a systematic review and a meta-analysis. Br J Anaesth. 2014 Jun;112(6):991-1004. doi: 10.1093/bja/aeu137. PMID 24829420
- [Background] Savage SR. Long-term opioid therapy: assessment of consequences and risks. J Pain Symptom Manage. 1996 May;11(5):274-86. doi: 10.1016/0885-3924(95)00202-2. PMID 8636626
- [Background] Chou R, Turner JA, Devine EB, Hansen RN, Sullivan SD, Blazina I, Dana T, Bougatsos C, Deyo RA. The effectiveness and risks of long-term opioid therapy for chronic pain: a systematic review for a National Institutes of Health Pathways to Prevention Workshop. Ann Intern Med. 2015 Feb 17;162(4):276-86. doi: 10.7326/M14-2559. PMID 25581257
- [Background] Katz J, Seltzer Z. Transition from acute to chronic postsurgical pain: risk factors and protective factors. Expert Rev Neurother. 2009 May;9(5):723-44. doi: 10.1586/ern.09.20. PMID 19402781
- [Background] Clarke H, Soneji N, Ko DT, Yun L, Wijeysundera DN. Rates and risk factors for prolonged opioid use after major surgery: population based cohort study. BMJ. 2014 Feb 11;348:g1251. doi: 10.1136/bmj.g1251. PMID 24519537
- [Background] Sun EC, Dixit A, Humphreys K, Darnall BD, Baker LC, Mackey S. Association between concurrent use of prescription opioids and benzodiazepines and overdose: retrospective analysis. BMJ. 2017 Mar 14;356:j760. doi: 10.1136/bmj.j760. PMID 28292769
- [Background] Katz J, Weinrib A, Fashler SR, Katznelzon R, Shah BR, Ladak SS, Jiang J, Li Q, McMillan K, Santa Mina D, Wentlandt K, McRae K, Tamir D, Lyn S, de Perrot M, Rao V, Grant D, Roche-Nagle G, Cleary SP, Hofer SO, Gilbert R, Wijeysundera D, Ritvo P, Janmohamed T, O'Leary G, Clarke H. The Toronto General Hospital Transitional Pain Service: development and implementation of a multidisciplinary program to prevent chronic postsurgical pain. J Pain Res. 2015 Oct 12;8:695-702. doi: 10.2147/JPR.S91924. eCollection 2015. PMID 26508886
- [Background] Weinrib AZ, Burns LC, Mu A, Azam MA, Ladak SS, McRae K, Katznelson R, Azargive S, Tran C, Katz J, Clarke H. A case report on the treatment of complex chronic pain and opioid dependence by a multidisciplinary transitional pain service using the ACT Matrix and buprenorphine/naloxone. J Pain Res. 2017 Mar 27;10:747-755. doi: 10.2147/JPR.S124566. eCollection 2017. PMID 28392713
- [Background] Tan G, Jensen MP, Thornby JI, Shanti BF. Validation of the Brief Pain Inventory for chronic nonmalignant pain. J Pain. 2004 Mar;5(2):133-7. doi: 10.1016/j.jpain.2003.12.005. PMID 15042521
- [Background] Rampakakis E, Ste-Marie PA, Sampalis JS, Karellis A, Shir Y, Fitzcharles MA. Real-life assessment of the validity of patient global impression of change in fibromyalgia. RMD Open. 2015 Sep 14;1(1):e000146. doi: 10.1136/rmdopen-2015-000146. eCollection 2015. PMID 26535150
- [Background] Portenoy R. Development and testing of a neuropathic pain screening questionnaire: ID Pain. Curr Med Res Opin. 2006 Aug;22(8):1555-65. doi: 10.1185/030079906X115702. PMID 16870080
- [Background] Dworkin RH, Turk DC, Wyrwich KW, Beaton D, Cleeland CS, Farrar JT, Haythornthwaite JA, Jensen MP, Kerns RD, Ader DN, Brandenburg N, Burke LB, Cella D, Chandler J, Cowan P, Dimitrova R, Dionne R, Hertz S, Jadad AR, Katz NP, Kehlet H, Kramer LD, Manning DC, McCormick C, McDermott MP, McQuay HJ, Patel S, Porter L, Quessy S, Rappaport BA, Rauschkolb C, Revicki DA, Rothman M, Schmader KE, Stacey BR, Stauffer JW, von Stein T, White RE, Witter J, Zavisic S. Interpreting the clinical importance of treatment outcomes in chronic pain clinical trials: IMMPACT recommendations. J Pain. 2008 Feb;9(2):105-21. doi: 10.1016/j.jpain.2007.09.005. Epub 2007 Dec 11. PMID 18055266
- [Background] Lowe B, Wahl I, Rose M, Spitzer C, Glaesmer H, Wingenfeld K, Schneider A, Brahler E. A 4-item measure of depression and anxiety: validation and standardization of the Patient Health Questionnaire-4 (PHQ-4) in the general population. J Affect Disord. 2010 Apr;122(1-2):86-95. doi: 10.1016/j.jad.2009.06.019. Epub 2009 Jul 17. PMID 19616305
- [Background] Darnall BD, Sturgeon JA, Cook KF, Taub CJ, Roy A, Burns JW, Sullivan M, Mackey SC. Development and Validation of a Daily Pain Catastrophizing Scale. J Pain. 2017 Sep;18(9):1139-1149. doi: 10.1016/j.jpain.2017.05.003. Epub 2017 May 19. PMID 28528981
- [Background] Wicksell RK, Renofalt J, Olsson GL, Bond FW, Melin L. Avoidance and cognitive fusion--central components in pain related disability? Development and preliminary validation of the Psychological Inflexibility in Pain Scale (PIPS). Eur J Pain. 2008 May;12(4):491-500. doi: 10.1016/j.ejpain.2007.08.003. Epub 2007 Sep 20. PMID 17884643
- [Background] Chapman SL, Jamison RN, Sanders SH. Treatment Helpfulness Questionnaire: a measure of patient satisfaction with treatment modalities provided in chronic pain management programs. Pain. 1996 Dec;68(2-3):349-61. doi: 10.1016/s0304-3959(96)03217-4. PMID 9121824